CLINICAL TRIAL: NCT06284278
Title: Comparison of Diaphragmatic Breathing Exercise and Pelvic Stabilization Exercise in Postpartum Women With Pregnancy-related Pelvic Girdle Pain: A Real-time Telehealth-based Intervention
Brief Title: Telehealth: Diaphragmatic vs. Pelvic Exercise in Postpartum Pregnancy-related Pelvic Girdle Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: YI-JU TSAI (Other)
Responsible Party: Sponsor-Investigator, YI-JU TSAI, professor, National Cheng Kung University
Organization: National Cheng Kung University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCKU_PPGP_diaphragm
Record Dates: First submitted 2023-09-19; First posted 2024-02-28 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Postpartum; Pregnancy Related; Pelvic Girdle Pain
MeSH Terms: conditions — Pelvic Girdle Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diaphragmatic breathing exercise group (Experimental): Diaphragmatic breathing exercise through telehealth
  Interventions: Other: Diaphragmatic breathing retraining; Other: pelvic anatomy education
- Pelvic stabilization exercise group (Active Comparator): Pelvic stabilization exercise through telehealth
  Interventions: Other: Pelvic stabilization exercise; Other: pelvic anatomy education

INTERVENTIONS:
Other: Diaphragmatic breathing retraining — 8 weeks diaphragmatic breathing training
  Arms: Diaphragmatic breathing exercise group
Other: Pelvic stabilization exercise — 8 weeks pelvic stabilization exercise training
  Arms: Pelvic stabilization exercise group
Other: pelvic anatomy education — pelvic anatomy education

SUMMARY:
The goal of this interventional study is to compare investigate the short-term and long-term effects of 8-week real-time telehealth-based diaphragmatic breathing exercise and pelvic stabilization exercise on pain, disability, and quality of life in postpartum women with pregnancy-related pelvic girdle pain.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-65 years
* Postpartum ≥ 3 months
* Pain located in sacroiliac joints (i.e., pain located between the posterior iliac crest and gluteal fold)
* Pregnancy-related cause of pelvic pain that pain occurs during pregnancy or after delivery (i.e., not traumatic or degenerative cause)
* At least 2 positive findings of 6 pain provocation tests for pelvic pain
* Score of Active Straight Leg Rise (ASLR) test > 0

Exclusion Criteria:

* being pregnant or actively trying to get pregnant
* having known causes of pelvic girdle pain, such as fractures and rheumatism
* having undergone lumbar, pelvic, gynecologic or obstetric surgery
* having current neurological symptoms and signs in lower extremities such as lumbar radiculopathy and myelopathy
* having cancer
* having cardiovascular disease
* being diagnosed as having a psychiatric disease
* active infection or infectious disease in the pelvis or abdomen
* having experience with structured and supervised core or trunk exercise training programs.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Muscle function measures of lumbopelvic muscles | Change from baseline to 8 weeks
  Ultrasonography image for muscle thickness of trunk and back muscles during rest and during active straight leg raise.
  Ultrasonography image for bladder displacement for pelvic floor muscles during rest,maximum contraction and during active straight leg raise
Diaphragm thickness | Change from baseline to 8 weeks
  Ultrasonography image for diaphragm thickness during maximum inspiration and expiration (B mode)
Diaphragm mobility | Change from baseline to 8 weeks
  Ultrasonography image for mobility during maximum inspiration and expiration (M mode)
Diaphragm strength | Change from baseline to 8 weeks
  Ultrasonography image for diaphragm strength during maximal sniff and expiration (M mode). The slope achieved (mm/sec) during the diaphragmatic excursion is used to calculate the velocity of the diaphragmatic contraction
Mechanical Property of Thoracolumbar Fascia | Change from baseline to 8 weeks
  The biomechanical and viscoelastic properties of the muscles will be measured using a non-invasive myometer. It automatically calculate and provide the biomechanical and viscoelastic properties of stiffness, frequency, decrement, and stress relaxation time that offer the information of tone, elasticity, stiffness and stress relaxation time of the tested tissue.
Functional performance of ASLR fatigue task | Change from baseline to 8 weeks
  Participants lifted the heel of the test leg to 20 cm for as long as possible. Participants were required to maintain pressure in the cuff beneath their back as close to 40 mm Hg as possible. Visual feedback of cuff pressure was provided throughout the task, but no instruction was given on how to affect cuff pressure. Task failure was defi ned as an inability to maintain heel height 10 cm or more off the plinth and/or a change in cuff pressure of 20 mm Hg or more.
Functional performance of timed up and go test | Change from baseline to 8 weeks
  Test instructions were given in Norwegian. Translated into English, the instructions were as follows: 'After "ready, set, go" stand up, walk as fast as you can until you cross the white line, turn around, and walk back to the chair and sit down again'. The white line was positioned 3m from the patient's starting position.
  'After "ready, set, go" stand up, walk as fast as you can until you cross the white line, turn around, and walk back to the chair and sit down again'. The white line was positioned 3m from the patient's starting position.
Functional performance of 6m timed walk test | Change from baseline to 8 weeks
  Subjects commenced the test in standing with their toes up against the tape marker. Test instructions translated into English were as follows: 'After "ready, set, go", walk as fast as you can up to the last white line without stopping or speaking along the way'. Performances were timed (to the nearest 100th of a second) between the 2m and 8m markers and later converted into speed in metres per second.
pain intensity measure of Numeric Rating Scale (NRS) | Change from baseline to 8 weeks
  Numeric Rating Scale (NRS) is a self-reported instrument assessing average pain intensity in currently. Possible score range from 0 (no pain) to 10 (worst possible pain).
Disability Level: measure of pelvic girdle questionnaire(PGQ) | Change from baseline to 8 weeks
  pelvic girdle questionnaire(PGQ) is a self-reported instrument assessing pelvic girdle pain intensity in currently. Questionnaire consisting of 20 activity items and 5 symptom items on a 4-point response scale. Possible score range from 0 (no pain) to 100 (worst possible pain).
Health-related Quality of Life: Short Form-36 (SF36) | Change from baseline to 8 weeks
  SF-36 include 36 questions constructing into 8 domains (i.e., physical functioning, physical role, bodily pain, general health, vitality, social functioning, emotional role, and mental health). The scores of physical and mental components and total are ranged from 0 to 100, with higher scores representing better quality of life
Fear Avoidance Belief: Tampa Scale of Kinesiophobia | Change from baseline to 8 weeks
  Fear of movement, fear of physical activity, and fear avoidance will be assessed using the Tampa scale of kinesiophobia (TSK). The TSK is 17-items questionnaire, where patients rate their agreement using 4-points scale. It consists of two subscales including activity avoidance to reflect the activity that may result in an increase in pain or cause injury, and somatic focus to reflect the beliefs and underlying serious conditions
Self-Efficacy: Pain Self-efficacy Questionnaire | Change from baseline to 8 weeks
  The pain self-efficacy questionnaire (PSEQ) is a 10-item questionnaire, where patients rate their confidence from 0 points (not at all confident) to 6 points (completely confident). Total scores of the PSEQ is 60 points and a higher score indicates more self-efficacy
Parenting Stress Level: Parenting Stress Index-Short Form (PSI-SF) | Change from baseline to 8 weeks
  The PSI-SF is a self-reported questionnaire that consists of 36 items to assess stress related to three aspects including parent-child relationship, parental distress, and difficulties in the parent-child interaction. The subscales for parental distress, parent-child dysfunctional interaction and difficult child, as well as the total stress scale are rated from 1 (strongly disagree) to 5 (strongly agree). The higher the score indicates the greater the stress.
Self-perceived Change: Global Rating of Change Scale (GROC) | Change from baseline to 8 weeks
  The GROC rates perceived "overall change" on a 15-point Likert scale, with 7 (labeled "worse") on the left, +7 (labeled "better") on the right, and 0 in the middle (labeled "no change") compared to the baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University, Tainan, Taiwan